CLINICAL TRIAL: NCT05934266
Title: Impact of Mesh Fixation With Tissue Adhesive on Open Inguinal Hernia Repair
Brief Title: Impact of Mesh Fixation With Tissue Adhesive
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario de Móstoles (Other)
Responsible Party: Principal Investigator, Justyna Drewniak Jakubowska, Surgeon, Hospital Universitario de Móstoles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUMostoles
Record Dates: First submitted 2023-06-12; First posted 2023-07-06 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Groin Hernia; Hernia, Inguinal; Postoperative Pain; Neuropathic Pain
Keywords: hernioplasty; mesh fixation; n-hexyl cyanoacrylate; groin hernia; postoperative pain
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tissue adhesive (Experimental): Group of 80 patients in which mesh fixation is done using cyanoacrylate glue
  Interventions: Device: Use of n-hexyl cyanoacrylate for mesh fixation
- Standard suture (No Intervention): Group of 80 patients who undergo hernioplasty with standard suture

INTERVENTIONS:
Device: Use of n-hexyl cyanoacrylate for mesh fixation — Mesh fixation with tissue adhesive (n-hexyl cyanoacrylate) in open hernia repair
  Arms: Tissue adhesive

SUMMARY:
Randomized controlled trial on mesh fixation using cyanoacrylate glue compared to standard suture in open inguinal hernia repair.

DETAILED DESCRIPTION:
Hernioplasty with suture-fixed mesh is the standard technique for the treatment of inguinal hernia, one of the most frequent pathologies in the Surgery Service. Despite its good results in terms of recurrences, it is currently under review due to the incidence of chronic postoperative pain. Up to half of the patients report some type of pain at one year of follow-up, and 15% report moderate-severe pain.

The objective of the study is to analyze whether the use of tissue adhesive (n-hexyl cyanoacrylate 0.5 ml) for mesh fixation in patients undergoing scheduled open inguinal hernioplasty results in a better postoperative evolution, with less chronic pain and less demand for analgesia, compared with a control group of patients who undergo the same surgical intervention with standard suture repair.

ELIGIBILITY:
Inclusion Criteria:

* Elective open inguinal hernioplasty in patients over 18 years old

Exclusion Criteria:

* Patient refusal
* Laparoscopic surgery
* Reintervention surgery
* Urgent surgery
* Cyanoacrylate allergy
* Administration of intraoperative local anesthetics
* Comorbidities that may affect the requirements of analgesics, such as degenerative arthropathies, fibromyalgia, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain assessed by visual numeric scale | 6 months
  Values come from 0 to 10, where 0 means no pain and 10 means the worst imaginable pain.
Postoperative administration of analgesics | 6 months
  Record of dose of analgesics needed: nonsteroidal anti-inflamatory drugs, opioid requirements, other analgesics requirements

SECONDARY OUTCOMES:
Hernia recurrence | 6 months
  Hernia recurrence rate after mesh fixation with tissue adhesive
Hematoma | 1 month
  Groin hematoma following hernioplasty with n-hexyl cyanoacrylate

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Móstoles, Móstoles, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code